CLINICAL TRIAL: NCT01274442
Title: A Case-control Study on the Impact of Genetic Polymorphisms on Dental Implant Loss.
Brief Title: Impact of Genetic Polymorphisms on Dental Implant Loss
Acronym: Polymorphism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010/771
Record Dates: First submitted 2011-01-10; First posted 2011-01-11 (Estimated); Last update posted 2022-12-29 (Actual); Status verified 2022-12

CONDITIONS: Patients Treated by Means of 1 or More Dental Implants
Keywords: dental implant
MeSH Terms: interventions — Immunologic Memory; Diagnosis, Oral; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CONTROL: no dental implants lost (Active Comparator): Group of patients who received an implant during a dental implant surgery in the University Hospital in Ghent in 2004-2007, who did not lose their implants.
  Interventions: Other: anamnesis; Procedure: oral examination; Procedure: Blood sample
- CASE: patients lost one or more implants (Experimental): Group of patients who received an implant during a dental implant surgery in the University Hospital in Ghent in 2004-2007, but who lost one or more implants.
  Interventions: Other: anamnesis; Procedure: oral examination; Procedure: Blood sample

INTERVENTIONS:
Other: anamnesis — To update the anamnesis.
Procedure: oral examination — A brief clinical oral examination will be performed.
Procedure: Blood sample — A blood sample will be taken to identify relevant genetic polymorphisms.

SUMMARY:
Patients that may participate in this case-control study underwent dental implant surgery in the University Hospital in Ghent in 2004-2007.

According to one of our recent papers based on this patient group, 34/461 patients lost one or more implants. The goal is to invite these 34 patients, to update the anamnesis, to perform a brief clinical oral examination and to have a blood sample. The latter is necessary to identify relevant genetic polymorphisms of the patient that are associated with implant loss. Among the remaining patients that did not lose implants, another 34 'controls' will be invited for the same examinations.

ELIGIBILITY:
Inclusion Criteria:

* Dental implant surgery in the University Hospital in Ghent in 2004-2007.
* Case: dental implant loss
* Control: no dental implant loss

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-06-01 (Actual); Primary Completion 2013-08-05 (Actual); Study Completion 2013-08-05 (Actual)

PRIMARY OUTCOMES:
genetic polymorphisms associated with implant loss | after 3 to 6 years
  Identification of genetic polymorphisms that are associated with implant loss. It concerns only one evaluation (1 blood sample).

CONTACTS AND LOCATIONS:
Overall Officials: Hugo De Bruyn, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Related Info — http://www.uzgent.be